CLINICAL TRIAL: NCT03078959
Title: The Prognostic Value of the Expression of Programmed Death Ligand 1 (PD-L1) in Early Stage Non-small-cell Lung Cancer
Brief Title: Prognostic Value of PD-L1 in NSCLC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondazione Ricerca Traslazionale (Other)
Responsible Party: Sponsor
Other Study IDs: L3P1490
Record Dates: First submitted 2017-03-03; First posted 2017-03-14 (Actual); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Immunohistochemistry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Formalin fixed paraffin embedded specimen were collected from 350 patients who underwent surgical resection of early stage NSCLC. Tumors samples were included in a tissue microarray.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: immunohistochemistry — Samples will be stained using the SP263 antibody clone against PD-L1

SUMMARY:
This is an observational retrospective study. The primary objective is to investigate the expression and potential prognostic role of Programmed Death Ligand 1 (PD-L1) in tumor samples from 350 patients with early stage treatment-naive non-small-cell lung cancer (NSCLC).

Tissue samples were embedded in a tissue microarray. PD-L1 will be studied by immunohistochemistry using the SP263 antibody. Stained samples will be evaluated independently by two operators. A tumor will be defined as positive when = or >50% of tumor cells express the ligand.

The investigators will investigate the relationship between PD-L1 protein expression and overall survival and other clinical characteristics with appropriate statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Early stage treatment-naive NSCLC

Exclusion Criteria:

* Received any pre-surgical treatment
* no OS data available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 350 patients with stagi I-III NSCLC
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2017-03-30 (Estimated); Study Completion 2017-04-15 (Estimated)

PRIMARY OUTCOMES:
Expression | 15 days
  The study will investigate PD-L1 protein expression by immunohistochemistry in tumor samples from early stage NSCLC
Prognostic value | 15 days
  The correlation between PD-L1 protein expression by immunohistochemistry and overall survival will be studied

IPD SHARING:
Plan to Share IPD: No